CLINICAL TRIAL: NCT05295875
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled and Parallel Group 48-Week Study to Evaluate the Efficacy and Safety of ALT-801 in the Treatment of Obesity (MOMENTUM Trial)
Brief Title: Efficacy and Safety of ALT-801 in the Treatment of Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-801-211
Record Dates: First submitted 2022-02-07; First posted 2022-03-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Obesity/Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — ALT-801

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALT-801 Dose Level 1 (Experimental)
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 2 (Experimental)
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 3 (Experimental)
  Interventions: Drug: ALT-801
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALT-801 — Injected subcutaneously (SC)
  Arms: ALT-801 Dose Level 1; ALT-801 Dose Level 2; ALT-801 Dose Level 3
Other: Placebo — Injected subcutaneously (SC)
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ALT-801 once-weekly versus placebo as an adjunct to a reduced-calorie diet and increased physical activity in patients with obesity/overweight.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed prior to entry into the study
* Male or female age 18 to 75 years, inclusive
* Body mass index (BMI) ≥ 30 kg/m2 or BMI ≥ 27 kg/m2 combined with at least one obesity-related comorbidity
* At least one unsuccessful weight loss attempt per investigator judgement
* Agreement to comply with the study-required life-style intervention and treatment during the full duration of the study
* Female subjects of childbearing potential who are not pregnant or breastfeeding, do not plan to become pregnant during the study, and agree to use effective birth control

Exclusion Criteria:

* Weight gain or loss > 5% in the 3 months prior to randomization or >10% in the 6 months prior to screening
* Diabetes and related conditions:

  1. History or clinical evidence of diabetes mellitus of any type, including Type 1, Type 2, or mature onset diabetes of the young (MODY)
  2. HbA1c > 6.5%, fasting glucose ≥ 126 mg/dL (6.9 mmol/L), and/or random glucose of ≥ 200 mg/dL (11.0mmol/L) at screening
* Obesity and related conditions:

  1. Obesity induced by known genetic causes or endocrine disorders (eg, Cushing Syndrome, inadequately treated hypothyroidism, defined as thyroid-stimulating hormone [TSH] > 6 mIU/L)
  2. History of bariatric surgery or other surgical treatment for obesity (eg, gastric banding, gastric bypass), or planned surgery or surgical treatment during the study. Liposuction and/or abdominoplasty performed >1 year before screening is allowed. Endoscopically placed intragastric balloons will be allowed if removed > 1 year before screening.
* Gastrointestinal conditions:

  1. History of acute or chronic pancreatitis within 1 year (365 days) before screening
  2. History of or acute significant gastrointestinal (GI) disorder (eg, peptic ulcers, severe gastroesophageal reflux disease [GERD],
  3. History of GI surgery, including cholecystectomy and antrectomy. Surgery for appendicitis and small bowel resection >20cm is acceptable.
  4. History of inflammatory bowel disease, celiac disease or any medical condition or surgery that could affect gastric emptying, stool frequency or stool consistency. (Irritable bowel syndrome is permitted provided that bowel frequency and consistency are normal off treatment.)
* Mental health conditions:

  1. Untreated depressive disorder, defined as a Patient Health Questionaire-9 (PHQ-9) score of ≥ 15 at screening
  2. Suicide ideation, defined as type 4 or 5 on the Columbia-Suicide Severity Rating Scale(C-SSRS) at screening, lifelong history of a suicide attempt, or suicidal behavior within 30 days before screening
  3. Other severe psychiatric disorder (eg, schizophrenia, bipolar disorder)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in body weight percentage | Baseline to Week 48

SECONDARY OUTCOMES:
Percent proportion of subjects with weight loss of greater than or equal to 5%, 10%, and 15% | Baseline to Week 48
Change from baseline in lipids | Baseline to Week 48
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Baseline to Week 48
Changes from baseline in Fasting Glucose | Baseline to Week 48
Changes from baseline in Hemoglobin A1c | Baseline to Week 48
Changes from baseline in Homeostatic Marker Assessment for Insulin Resistance (HOMA-IR) | Baseline to Week 48
Changes from baseline in: a) Systolic blood pressure, b) Diastolic blood pressure | Baseline to Week 48
Change from baseline in proportion of patients using antihypertensive medications | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Browne, MD, Study Director — Altimmune, Inc.
Locations (31):
- United States (31):
  - Altimmune CTM, Birmingham, Alabama
  - Altimmune CTM, Mesa, Arizona
  - Altimmune CTM, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Altimmune CTM, Montclair, California
  - Altimmune CTM, Santa Barbara, California
  - Altimmune CTM, Boca Raton, Florida
  - Altimmune CTM, Clearwater, Florida
  - Altimmune CTM, Fort Myers, Florida
  - Altimmune CTM, Jacksonville, Florida
  - Altimmune CTM, Port Orange, Florida
  - Altimmune CTM, Sunrise, Florida
  - Altimmune CTM, Savannah, Georgia
  - Altimmune CTM, Evanston, Illinois
  - Altimmune CTM, Indianapolis, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Altimmune CTM, Louisville, Kentucky
  - Altimmune CTM, Baton Rouge, Louisiana
  - Altimmune CTM, New Orleans, Louisiana
  - Altimmune CTM, Kansas City, Missouri
  - Altimmune CTM, Butte, Montana
  - Altimmune CTM, Berlin, New Jersey
  - Altimmune CTM, New York, New York
  - Cornell University, Joan and Sanford Weill Medical College, New York, New York
  - Altimmune CTM, Cincinnati, Ohio
  - Altimmune CTM, Philadelphia, Pennsylvania
  - Altimmune CTM, Knoxville, Tennessee
  - Altimmune CTM, Austin, Texas
  - Altimmune CTM, Bellaire, Texas
  - Altimmune CTM, San Antonio, Texas
  - Altimmune CTM, St. George, Utah